CLINICAL TRIAL: NCT01989819
Title: Primary Sjögren Syndrome
Acronym: NeuroSenSS
Status: Completed | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: I10 023
Record Dates: First submitted 2013-11-06; First posted 2013-11-21 (Estimated); Last update posted 2019-01-11 (Actual); Status verified 2016-06

CONDITIONS: Primary Sjögren's Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- patients with Sjögren's syndrome: A skin biopsy will be performed in patients
  Interventions: Other: skin biopsy
- control group: A skin biopsy will be performed in control group
  Interventions: Other: skin biopsy
- non auto-immune small fiber neuropathies

INTERVENTIONS:
Other: skin biopsy
  Groups: control group; patients with Sjögren's syndrome

SUMMARY:
Primary Sjögren syndrome (pSS) is an inflammatory, autoimmune, multiorgan disease often involving the central and peripheral nervous systems. Fifteen to twenty percent of patients with the primary Sjögren's syndrome have neurological complications involving the peripheral nervous system. Although some patients have large fiber neuropathy, around forty percent of patients with Sjögren's syndrome experience neuropathic pain with normal electrodiagnostic studies. Although these patients may be diagnosed with fibromyalgia or depressive symptoms, some have been shown to have small fiber neuropathy (SFN). A recent study proved that more than 90% of pSS patients with such neuropathic pain have SFN {Fauchais, 2010 #188}.

The aim of this study will be to investigate the occurrence of small fiber neuropathy in patients with pSS and neuropathic pain with normal electromyographic studies and to determine the existence of a conjoint local inflammatory process mediated by cellular, cytokinic or auto-antibody response. Quantification of epidermal nerve fiber density after skin biopsy is a valuable tool to diagnose small fiber neuropathy and the method has been widely validated. A skin biopsy will be performed in patients and control and will allow quantification of small fiber density in skin sample along with measurement of sweat gland innervation. Moreover, pathophysiological studies will be carried on in order to evaluate the causal relationship between cellular and humoral inflammation and small fiberneuropathy.

Recent studies have pointed out the inconstant efficacy of both corticosteroid and immunosuppressive drugs in pSS-related SFN. Dissecting the molecular mechanisms of small fiber neuropathy in these patients may help designing new therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pSS according to revised European criteria and exhibiting neuropathic pain without any electromyographic abnormality will be included (Group I).
* Age of entry into the study ≥ 18 yrs (both groups).
* Affiliated or profit patient of a social security system (both groups).
* Informed consent signed up (both groups).

Exclusion Criteria:

* Chronic alcoholism
* Type I or type II diabetes
* Peripheral neuropathy unrelated to pSS complications
* Coagulation disease
* Previous allergy to xylocaine, lidocaine, prilocaine or ricin oil
* Porphyria, methemoglobinemia
* Patients under measure of maintenance of justice.
* Patients unable to understand or to participate to the study.
* Child and major patients making the object of a measure of lawful protection.
* Patients deprived of freedom.
* Pregnant, nursing women.
* Participation in biomedical research within one month prior to inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Sjögren's syndrome
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the cutaneous lymphocytic infiltration | 1 year

SECONDARY OUTCOMES:
Cutaneous infiltration T, B and Th17 | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Laure FAUCHAIS, MD, Principal Investigator — University Hospital, Limoges
Locations (7):
- France (7):
  - CH d'Albi, Albi
  - CHU Bordeaux, Bordeaux
  - CH de Brive, Brive-la-Gaillarde
  - CHU de Lille, Lille
  - University Hospital, Limoges, Limoges
  - CH de Rodez, Rodez
  - CHU Toulouse, Toulouse